CLINICAL TRIAL: NCT05304117
Title: Culturally Tailoring an Advance Care Planning Intervention for American Indians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Carolina University (Other)
Collaborators: Pacific Institute for Research and Evaluation (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Elizabeth Anderson, Assistant Professor of Social Work, Western Carolina University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1685879-1; 1R21NR019910-01 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-03-31 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Advance Care Planning
Keywords: American Indian; Advance Care Planning; Serious illness; end-of-life care
MeSH Terms: interventions — Advance Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance Care Planning Experimental (Experimental): Community Information Session on advance care planning and private one-on-one Sharing Session about advance care planning.
  Interventions: Behavioral: Advance Care Planning
- Advance Care Planning Waitlist (Other): Waitlist Group- Baseline control measures will be collected at consent and again 3-6 months later before attending a Community Information Session on advance care planning and an one-on-one Sharing Session about Advance Care Planning. Data will be collected again 8 weeks after the intervention.
  Interventions: Behavioral: Advance Care Planning

INTERVENTIONS:
Behavioral: Advance Care Planning — Community Information Session and Private Sharing Session with trained social worker

SUMMARY:
This project has three specific aims: (1) culturally tailor the content of the Make Your Wishes about You (MY WAY) ACP curriculum and guide for one American Indian tribe; (2) assess the feasibility of the culturally-tailored MY WAY ACP curriculum and patient education guide with the tribe; and (3) examine preliminary outcomes of the culturally-tailored MY WAY ACP curriculum and guide with 70 tribal members. Upon successful completion, it is expected that this project will develop a feasible culturally-tailored MY WAY that through a quasi-experimental waitlist design shows promise as an efficacious program with respect to self-efficacy, readiness, and ACP completion that increases facilitators and decreases barriers to ACP.

DETAILED DESCRIPTION:
Research Design. A quasi-experimental waitlist study design will be used to test the hypothesis that the intervention participants will experience increased ACP self-efficacy, readiness, and completion rates. It is also expected that the intervention participants will experience increased facilitators and decreased barriers to ACP. A control sample of waitlist participants will be used.

Based on the odds of completing an ACP indicated in previously implemented MY WAY interventions and using 90% power as a threshold, it is estimated that will be a need for at least an n = 60 to find effects. The intervention group, Cohort 1, will be those who participated in the first round of both the Community Educational Sessions and Sharing Sessions. The control group, Cohort 2, will be those who participated in the second round of both the Community Education Sessions and Sharing Sessions.

Measurement. Process Measures that are a part of the 9-item ACP Engagement Survey that includes measurement of self-efficacy and readiness, identified from Behavioral Change Theory, will be used. Self-efficacy and readiness subscales have Likert responses of "not at all, a little, somewhat, fairly, extremely" and have good reliability and discriminant validity. Barriers and Facilitators to ACP Questionnaire used in the MY WAY randomized controlled trial will be used. Pretest interviews with these measurements will be conducted by telephone or in person at the time of pre-registration for both cohorts by the Project Coordinator and team members.

Cohort 1 will be interviewed five times: Baseline pretest, Community Information Session Evaluation; Sharing Session Evaluation, 8 week-post test and 6 month post-test.

Cohort 2 will be interviewed five times: Baseline pretest, 2nd baseline control pretest, waitlist Community Information Session evaluation, and waitlist Sharing Session evaluation, 8 week post test.

The first interview at registration will serve as baseline for the waitlist group, Cohort 2. Cohort 2 will be contacted again approximately 6 months later and two-weeks prior to the second Community Education Session to remind them of their registration and to re-interview them for their intervention pretest. Posttest interviews will also be conducted by the Project Coordinator eight weeks post Sharing Session for both groups to capture ACP self-efficacy, readiness, and completion rates.

Statistical Analyses. Demographic characteristics will be examined using descriptive statistics (frequencies, measures of central tendency, measures of variation) and stratified analyses (e.g., delineating measures by demographics, attendance, ACP agreement etc.) to examine the association between demographics and program outcomes. ACP Engagement and the Barriers and Facilitators to ACP Questionnaire (ACP measures) will be compared between those who do and do not engage in Sharing Sessions and between Cohort 1 and Cohort 2. The tribal community as well as location of Community Education Session will be included in all analyses as nested participant variables to ensure that differences between tribal communities and education delivery do not significantly change results. To account for these nested variables, hierarchical linear modeling or a similar method will be used in comparison analyses. It is likely that there will be significant attrition from Community Education Sessions to Sharing Sessions. A Heckman Selectivity analyses will be used to determine if there are differences between those who complete the full intervention and those who complete only baseline measures or Community Educational Sessions. Due to the nature of the study, there may also be attrition due to death. If there are differences in attrition, the inverse Mill's ratio will be used in all further analyses. Comparison of baseline measures from pre-registration interviews will serve to ensure that there are no significant differences between the cohorts.

After these preliminary analyses, change in Cohort 1's ACP measures can be compared to changes from baseline to the waitlist pretest measures from Cohort 2. Since Cohort 2 received no intervention in the first 6 months, the analysis will control for natural variations over time and any measures which show significantly larger change in Cohort 1 can be attributed to the intervention. Cohorts 1 and 2 can then be combined to examine intervention effects (i.e., change from pretest to posttest) in the full sample of participants who experienced the Sharing Sessions; baseline results for Cohort 1 will be combined with waitlist pretest results for Cohort 2 and compared to the combined group of 70 Sharing Sessions' posttests. Finally, the combined cohorts will be compared to a subsample of matched participants who experienced the Community Education Sessions only to determine how each step in MY WAY affects the outcome ACP measures.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* either enrolled member or spouse of enrolled member in tribal service area
* Member of another American Indian/Alaskan Native tribe
* English fluency
* Resides in the tribal service area.

Exclusion Criteria:

• Cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R T Goins, PhD, Principal Investigator — Western Carolina University
Locations (1):
- Western Carolina University, Asheville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schweinhart A, Goins RT, Anderson E. Results of a Culturally Tailored Advance Care Planning Intervention for American Indian Peoples: A Quasi-Experimental Waitlist-Controlled Trial. Innov Aging. 2025 May 6;9(6):igaf041. doi: 10.1093/geroni/igaf041. eCollection 2025. PMID 40520470
- [Derived] Anderson E, Goins RT, Haozous EA, Schweinhart A. Testing a Culturally Tailored Advance Care Planning Intervention (MY WAY) for an American Indian Tribe: Protocol for a Quasi-Experimental Waitlist Control Design. JMIR Res Protoc. 2023 Dec 29;12:e50654. doi: 10.2196/50654. PMID 38157237

RESULTS

PARTICIPANT FLOW:
Groups:
- Advance Care Planning Waitlist: Waitlist Group- Baseline control measures will be collected at the same time as Cohort 1 completes their pretest. Six Months after Cohort 1, participants will be pretested again before attending a Community Information Session on advance care planning and an one-on-one Sharing Session about Advance Care Planning.
  Advance Care Planning: Community Information Session and Private Sharing Session with trained social worker
Period: Overall Study
Arm/Group | Advance Care Planning Experimental | Advance Care Planning Waitlist
Started | 114 | 41
Completed | 105 | 41
Not Completed | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advance Care Planning Experimental | Advance Care Planning Waitlist | Total
Number analyzed (Participants) | 114 | 41 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 13 | 58
  >=65 years | 69 | 28 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.93 (16.7) | 68.3 (13.8) | 64.82 (15.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 28 | 109
  Male | 33 | 13 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 96 | 35 | 131
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 6 | 24
Region of Enrollment [Number; unit: participants]
  United States | 114 | 41 | 155
Advance Care Plans [Count of Participants; unit: Participants] | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Count of Self-Report of Advance Directive
Description: The proportion of participants who self-report advance directive completion.
Time Frame: Cohort 1 Experimental: Baseline and Post-test (week 8); Cohort 2 Waitlist: Baseline 1 and Baseline 2 (3-6 months after baseline and immediately before intervention); Cohort 2 Experimental; Baseline 1 and post-test (5-8 months after 1st baseline)
Measure: Count of Participants; unit: Participants
Groups:
- Advance Care Planning Experimental (Cohort 1): Community Information Session on advance care planning and private one-on-one Sharing Session about advance care planning.
  Advance Care Planning: Community Information Session and Private Sharing Session with trained social worker
- Advance Care Planning Waitlist (Cohort 2): Waitlist Group- Baseline control measures collected at consent, and again 3-6 months later before attending a Community Information Session on advance care planning and a one-on-one Sharing Session about Advance Care Planning. Data also collected 8 weeks post intervention.
Arm/Group | Advance Care Planning Experimental (Cohort 1) | Advance Care Planning Waitlist (Cohort 2)
Number analyzed (Participants) | 105 | 41
Participants
  Baseline | 10 | 5
  Cohort 1-8 weeks after intervention; Cohort 2- 3-6 months after baseline but before intervention | 67 | 6
  Cohort 1- 6 months after intervention; Cohort 2- 8 weeks after intervention | 67 | 29

2. Primary Outcome: Average Advance Care Planning -Engagement Readiness
Description: The mean ACP Readiness scores range from 1-6, with higher scores indicating greater readiness.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Advance Care Planning Experimental Group (Cohort 1): Participants in this arm had a baseline survey immediately before the intervention. Participants in this arm had a post-test survey 8 weeks after the intervention.
- Advance Care Planning Waitlist- Cohort 2: Participants in this arm had a baseline (control) survey and then were waitlisted for 3-6 months. The 2nd baseline was repeated at 3-6 months, before the intervention.
- Advance Care Planning Experimental Cohort 2: Participants in this arm had a baseline survey and then were waitlisted for the intervention for approximately 3-6 months, and were given a post-test 5-8 months after the 1st baseline (8 weeks after intervention).
Arm/Group | Advance Care Planning Experimental Group (Cohort 1) | Advance Care Planning Waitlist- Cohort 2 | Advance Care Planning Experimental Cohort 2
Number analyzed (Participants) | 91 | 41 | 37
score on a scale
  Baseline | 3.20 (1.01) | 3.26 (1.05) | 3.26 (1.05)
  post-test | 4.12 (0.80) | 3.56 (0.87) | 4.26 (0.76)

3. Primary Outcome: Average Advance Care Planning-Engagement Self-Efficacy
Description: The mean ACP Self-Efficacy scores range from 1-6, with higher scores indicating greater self-efficacy.
  not at all, a little, somewhat, fairly, extremely Higher scores indicate better outcomes.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Advance Care Planning Experimental (Cohort 1): Participants in this arm had a baseline survey immediately before the intervention. Participants in this arm had a post-test survey 8 weeks after the intervention.
- Advance Care Planning Waitlist (Cohort 2): Participants in this arm had a baseline (control) survey and then were waitlisted for 3-6 months. The 2nd baseline was repeated at 3-6 months, before the intervention.
- Advance Care Planning Experimental (Cohort 2): Participants in this arm had a baseline survey and then were waitlisted for the intervention for approximately 3-6 months, and were given a post-test 5-8 months after baseline (8 weeks after intervention).
Arm/Group | Advance Care Planning Experimental (Cohort 1) | Advance Care Planning Waitlist (Cohort 2) | Advance Care Planning Experimental (Cohort 2)
Number analyzed (Participants) | 91 | 41 | 37
score on a scale
  Baseline | 4.33 (0.93) | 4.28 (0.99) | 4.28 (0.99)
  8 weeks | 5.29 (0.85) | 4.84 (0.87) | 5.56 (0.42)

4. Secondary Outcome: Average Number of Barriers to Advance Care Planning
Description: The sum (0-8) ACP Barriers Score with higher scores indicating more barriers.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Advance Care Planning Experimental (Cohort 1): Participants in this arm had a baseline survey immediately before the intervention, and then again 8 weeks post intervention.
- Advance Care Planning Experimental (Cohort 2): Participants in this arm had a baseline survey and then were waitlisted for the intervention for approximately 3-6 months, and were given a post-test 5-8 months after 1st baseline (8 weeks post intervention).
Arm/Group | Advance Care Planning Experimental (Cohort 1) | Advance Care Planning Waitlist (Cohort 2) | Advance Care Planning Experimental (Cohort 2)
Number analyzed (Participants) | 91 | 41 | 37
score on a scale
  Baseline | 1.96 (1.93) | 2.39 (2.23) | 2.39 (2.23)
  Post-test | 1.44 (1.97) | 1.44 (1.6) | 1.11 (1.31)

5. Secondary Outcome: Average Number of Facilitators for Advance Care Planning
Description: The sum (0-8) of ACP Facilitators Score , with higher scores indicating more facilitators.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Advance Care Planning Experimental (Cohort 2): Participants in this arm had a baseline survey and then were waitlisted for the intervention for approximately 3-6 months, and were given a post-test 5-8 months after the 1st baseline (8 weeks following the intervention).
Arm/Group | Advance Care Planning Experimental (Cohort 1) | Advance Care Planning Waitlist (Cohort 2) | Advance Care Planning Experimental (Cohort 2)
Number analyzed (Participants) | 91 | 41 | 37
score on a scale
  Baseline | 5.65 (1.44) | 6.24 (1.2) | 6.24 (1.2)
  Post-test | 6.52 (1.43) | 5.95 (1.55) | 5.19 (1.27)

ADVERSE EVENTS:
Time Frame: Through study completion, up to 8 months.
Description: This intervention was voluntary and participants provided informed consent prior to enrollment. There is little data that suggests that advance care planning causes adverse effects. The intervention instructed participants that they could stop at any time. Support Stars and Project Coordinator worked closely with participants over time and were instructed to inform PIs of any potential adverse events, but none were noted. PI's learned of 3 participants deaths throughout the study, unrelated.
Arm/Group | Advance Care Planning Experimental | Advance Care Planning Waitlist
All-Cause Mortality (participants affected / at risk) | 3/105 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/41
Other Adverse Events (participants affected / at risk) | 0/105 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT05304117/Prot_SAP_000.pdf